CLINICAL TRIAL: NCT05748704
Title: Phase I / II Single Arm Study: Metabolic and Immunological Effects of a Modified Fasting Regimen in Cancer Patients
Brief Title: Metabolic and Immunological Effects of a Modified Fasting Regimen in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Alessio Nencioni, Principal Investigator, University of Genova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STMF
Record Dates: First submitted 2022-10-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: fasting; short-term modified fasting
MeSH Terms: conditions — Neoplasms; Fasting

STUDY DESIGN:
Intervention Model Description: STMF is a 5-day low-calorie and low-protein (totally plant-based) diet that involves a short-term modified fast.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-term modified fasting (Experimental): The STMF regimen consists of a low-calorie diet lasting five days and aimed at providing between 800 and 1,000 kcal/day (tentatively 10% carbohydrates, 15% proteins, 75% lipids).
  Interventions: Other: Short-term modified fasting

INTERVENTIONS:
Other: Short-term modified fasting — STMF regimen consists of a low-calorie diet aimed at providing 800-1,000 kcal/day, lasting five days and with the following composition: 10% carbohydrates, 15% proteins, 75% lipids. During the days of STMF, patients will be required to write down the foods consumed in a food diary in order to calculate calorie and nutrients intake. The STMF regimen will be administered tentatively on a monthly basis (depending on the therapeutic regimen the patient undergoes) and in any case no more frequently than once every three weeks.

SUMMARY:
This is a single-arm prospective pilot study assessing the metabolic and immunologic effects of a modified fasting regimen in cancer patients with different cancer types and concomitant anticancer treatment.

DETAILED DESCRIPTION:
A single-arm phase II clinical trial of a short-term modified fasting regimen (STMF) is proposed to be conducted in 100 patients with solid tumors who are candidates to receive active medical or radiotherapy treatment (or with medical treatment or radiotherapy already ongoing). Cancer treatment can be adjuvant or palliative. Patients with haematological tumors are also included. Enrolment is also foreseen for patients with haematological tumors who are not undergoing active treatment yet, but are followed with a watchful waiting approach (e.g. patients with low-risk B-CLL or low-risk follicular lymphoma). Finally, enrolment is also open to patients with relapsing forms of non-melanoma skin cancers (e.g. basalioma, epithelioma).

The primary endpoint of the study is to evaluate the effects of a STMF on the circulating levels of factors with pro- or anti-oncogenic activity (including insulin, IGF1, IGFBP1, IGFBP3 , leptin, adiponectin, IL-6, TNF-alpha, IL1beta), as well as the effect of STMF cycles on leukocyte subpopulations with a role in the control of tumor growth, such as regulatory T cells, the "myeloid-derived suppressor cells" (MDSC) as well as NK cells, and on stem cell pools (e.g. hematopoietic stem cells, endothelial stem cells, mesenchymal stem cells).

The STMF regimen that is applied is a 5-day low-calorie and low-protein diet. Patients undergo a medical exam/history collection and a nutritional assessment (body weight, handgrip strenght and bioimpedance measurement) at baseline and then at the visits that precede every cycle of STMF (i.e. once every three weeks or monthly, depending on the therapeutic regimen the patient is undergoing, and in any case no more frequently than once every three weeks - eg when combined with q21 chemotherapy regimens). Adverse events are recorded at each visit in accordance with NCI-CTCAE version 5.0. P

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Patients with solid or hematologic tumors undergoing active treatment (including chemotherapy regimens, hormone therapies, other molecularly targeted therapies - including kinase inhibitors, biologicals or inhibitors of immune checkpoints; patients in whom treatment is already ongoing are also eligible; patients with haematological malignancies who are managed by watchful waiting (e.g. low-risk B-CLL or follicular lymphoma) as well as patients with relapsing forms of non-melanoma skin cancer (basal or squamous cell carcinoma) are also eligible.
* ECOG performance status 0-1
* Adequate organ function
* BMI >21 kg/m2 (with possibility to also enroll patients with 18.5<BMI<21 based on the judgement of the treating physician)
* Low nutritional risk according to nutritional risk screening (NRS)

Exclusion Criteria:

* Age> 65 years [with the possibility to enroll from 65 to 75 years old patients if considered safe by the examining doctor
* Diabetes mellitus;
* BMI <18.5 kg/m2;
* Bio-impedance phase angle <5.0°;
* Medium/high nutritional risk according to NRS;
* Any metabolic disorder capable of affecting gluconeogenesis or the ability to adapt to periods of fasting;
* Ongoing treatment with other experimental therapies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Effects of the STMF on IGF1 and IGFBP1 | month 1-12
  IGF1 and IGFBP1 dosage (μg/l)
Effects of the STMF on IGFBP3 | month 1-12
  IGFBP1 dosage (mg/l)
Effects of the STMF on Interleukin-6 (IL-6), interleukin-1 beta (IL1-beta) and tumor necrosis factor-alpha (TNF-alpha) | month 1-12
  IL-6, IL-1beta and TNF-alpha dosage (pg/ml)
Effects of the STMF on insulin | month 1-12
  Insulin dosage (mLU/L)
Effects of the STMF on adiponectin | month 1-12
  Adiponectin dosage (μg/ml)
Effects of the STMF on leptin | month 1-12
  Leptin dosage (ng/ml)

SECONDARY OUTCOMES:
Percentage of prescribed diet consumed and intake of any extra food | 3 to 8 weeks depending on the patient's therapy
  It will be assessed using a food diary during 5 days of STMF and is defined as strict adherence to the diet; it is permitted a maximum consumption of 5 Kcal / kg of body weight of extra food on only one of the days of each cycle; or a maximum consumption of 2 Kcal / kg of body weight of extra food in two days of each cycle; or as the reduction of the number of days of the STMF from 5 to 3/4 at most once every three cycles.
Quantification of emergent adverse events | 3 to 8 weeks depending on the patient's therapy
  It will be assessed monitoring adverse events during STMF according to CTCAE 5.0.
Body Weight | 3 to 8 weeks depending on the patient's therapy
  Weight is used to calculate the BMI as weight (kg)/height (m2).
Effect of STMF on circulating tumor DNA | month 1-12
  It will be assessed by measuring circulating tumor DNA - ctDNA
Effect of the STMF on the intestinal microbiome | month 1-3
  It will be assessed by comparing fecal samples: the investigators are going to collect simples before and after the first and the third cycle. The analysis will be carried out through the analysis of the 16S rRNA present in the sample. The investigators will analyze if and how bacterial strains change in terms of quantity and quantity after cycles of fasting
Phase Angle (PA) | 3 to 8 weeks depending on the patient's therapy
  PA is a linear method of measuring the relationship between Electrical Resistance (Rz) and Reactance (Xc) both expressed in ohms (Ω). PA is detected by a Single Frequency Bioimpedance Analyzer (BIA 101®, Akern, Florence, Italy). Bioelectrical impedance measurements are subsequently processed with the Bodygram Plus® software (Akern, Florence, Italy). PA is an indicator of nutritional status
Handgrip strength | 3 to 8 weeks depending on the patient's therapy
  Handgrip strength is evaluated with the use of a dynamometer (T.K.K.5001 GRIP A Hand Grip Analogue Dynamometer, Takei, Japan).
Effect of cycles of STMF on leukocyte subpopulations | month 1-12
  To evaluate the potential impact of fasting on antitumor immune response, we will use multicolor flow cytometry to explore the frequency of myeloid and lymphocytic peripheral blood mononuclear cell (PBMC) populations, with a particular focus on natural killer (NK) cells (CD45+ CD3- CD56+ CD16+ DR+/-), B cells (CD3-CD45+ CD19+), T cells (CD3+ CD45+), NKT cells (CD45+ CD3+ CD56+ CD16+ DR+/-), helper T (Th) cells (CD3+ CD45+ CD4+ DR+/-), cytotoxic T (CTL) lymphocytes (CD3+ CD45+ CD8+ DR+/-), regulatory T (Treg) cells (CD3+ CD45+ CD8+/- CD4+/- CD127- CD25+), exhausted T cells (CD3+ CD45+ CD8+/- CD4+/- CD28-), activated and effector T cells (CD3+ CD45+ CD8+/- CD4+/- CD39+ CD25+ DR+).

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Nencioni, MD, Principal Investigator — Universita degli Studi di Genova
Locations (1):
- San Martino Hospital, Genova, Italy

IPD SHARING:
Plan to Share IPD: No